CLINICAL TRIAL: NCT02980991
Title: Pemetrexed and Platinum Use in the Neoadjuvant Setting for Resectable Stage II and IIIA Lung Adenocarcinoma
Brief Title: Pemetrexed and Platinum Use in the Neoadjuvant Setting for Resectable Stage II and IIIA Lung Adenocarcinoma (ECTOP-1002)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Director of Department of Thoracic Surgery, Shanghai Cancer Center, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCPOII
Record Dates: First submitted 2014-12-16; First posted 2016-12-02 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Lung Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Pemetrexed; Neoadjuvant Therapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant chemotherapy group (Experimental): Two cycles of pemetrexed and cisplatin given to patients before surgery
  Interventions: Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Pemetrexed — Two cycles of pemetrexed 500mg/m2 day 1, 21 days per cycle for patients before surgery
  Other Names: Neoadjuvant chemotherapy
Drug: Cisplatin — Two cycles of cisplatin 75mg/m2 day 1 (or 25mg/m2 day 1-3), 21 days per cycle for patients before surgery
  Other Names: Neoadjuvant chemotherapy

SUMMARY:
This is a clinical trial from Eastern Cooperative Thoracic Oncology Project (ECTOP), numbered as ECTOP-1002. The study is a prospective, single-center, open-label, single-armed, phase II clinical trial. The aim of the study is to evaluate the radiological response rate (RR) of 2 cycles of neoadjuvant chemotherapy with pemetrexed and cisplatin in patients with resectable stage II and IIIA lung adenocarcinoma.

DETAILED DESCRIPTION:
The study is a prospective, single-center, open-label, single-armed, phase II clinical trial. Clinical staging is determined according to the routine protocol, which include enhanced chest CT scans, brain MRI or CT, bone scintigraphy, abdominal ultrasonography and cardiopulmonary tests. PET/CT scan was optional. Preoperative diagnoses of lymph node metastasis were performed using enhanced chest CT or PET/CT. Preoperative pathological diagnosis is confirmed by electronic fiber bronchoscopic biopsy, CT-guided percutaneous lung puncture biopsy and endobronchial ultrasonography （EBUS/EUS） when necessary.

Patients are going to receive two cycles of pemetrexed 500mg/m2 day 1 and cisplatin 75mg/m2 day 1 (or 25mg/m2 day 1-3), 21 days per cycle. Treatment cycles are repeated every 21 days. Following two cycles of chemotherapy, the same radiological examination as baseline chest CT or PET/CT scans are repeated for tumor response evaluation. Radiographic response was recorded by Response Evaluation Criteria in Solid Tumors （RECIST 1.1）. Patients undergo complete resection between 2 and 6weeks following the last dose of chemotherapy. The surgical extents left to the discretion of the general thoracic surgeon. And lobectomy and pneumonectomy with mediastinal lymph node dissection are recommended. Two cycles of post-surgery pemetrexed/cisplatin treatment will be administrated subsequently.

The primary objective is to determine the radiological response rate (RR) of 2 cycles of neoadjuvant chemotherapy with pemetrexed and cisplatin in patients with resectable stage II and IIIA lung adenocarcinoma. The radiological response rate is measured 3 to 4 weeks after the second cycle of chemotherapy according to the RECIST criteria 1.1.

The secondary objectives are to determine the pathological response rate, safety, the clinical feasibility rate, the drug delivery, 2-year disease free survival (DFS) and 2-year overall survival (OS).The pathological response rate is investigated by determination of the type and extent of vital tumor tissue and tumor necroses as well as reactive alterations with foam cell reaction and fibrosis or scar formation on light microscopic evaluation of surgical resection specimens stained with H&E.The clinical feasibility is achieved if 1) no death due to cancer, toxicity or comorbidity,and 2) no toxicity events including Grade 4 neutropenia >7 days; febrile grade 3/4 neutropenia; grade 4 thrombocytopenia >7 days or any grade with bleeding; grade 3/4 nonhematologic toxicity related to chemotherapy (except nausea/vomiting/hair loss) are observed. The drug delivery is defined as the accomplishment of the chemotherapy.DFS is measured from the date of operation until the date of first progression or recurrence. OS is measured from the date of operation until the date of death from NSCLC or the date last seen alive.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent must be signed.
2. At least 18 years of age.
3. Histologically or cytologically diagnosed as lung adenocarcinoma.
4. Have measurable and clinical stage II-IIIA (excluding superior sulcus) disease eligible for surgery.
5. No previous systematic therapy or radiotherapy.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Have a predicted postresection forced expiratory volume in 1 second (FEV1) of ≧1.0 L.
8. Have adequate organ function including the following:

   Bone marrow: absolute neutrophil count (ANC) ≥1.5*109/L, platelets ≥100*109/L, hemoglobin ≥8 g/dL.

   Hepatic: bilirubin ≤1.5 ULN, alkaline phosphatase (AP), aspartate transaminase (AST), and alanine transaminase (ALT) ≤3.0 ULN.

   Renal: calculated creatinine clearance ≥45 mL/min (using the standard Cockcroft-Gault formula).
9. For women: must be surgically sterile, postmenopausal, or compliant with a medically approved contraceptive regimen during and for 3 months after the treatment period; must have negative serum or urine pregnancy test and must not be lactating. For men: must be surgically sterile, or compliant with a contraceptive regimen during and for 3 months after the treatment period.

Exclusion Criteria:

1. Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry or concurrent administration of any other anti-tumor therapy.
2. Clinically diagnosed as stage I or IIIB.
3. Have history of another malignancy within the last 5 years except cured carcinoma in-situ of uterine cervix, cured basal cell carcinoma of skin and superficial bladder tumors [Ta, Tis & T1].
4. Concurrent use of any other anti-cancer therapy during study treatment.
5. Any unstable systemic disease (including active infection, hepatic, renal or metabolic disease) or serious concomitant disorders that would compromise the safety of the patient, or compromise the patient's ability to complete the study, at the discretion of the investigator.
6. Significant cardiovascular event: congestive heart failure > New York Heart Association (NYHA) class 2; unstable angina, active CAD (myocardial infarction more than 1 year prior to study entry is allowed); serious cardiac arrhythmia requiring anti-arrythmic therapy (beta-blockers or digoxin are permitted) or uncontrolled hypertension.
7. Inability to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs) 2 days before, the day of, and 2 days after the dose of pemetrexed. If a patient is taking an NSAID (Cox-2 inhibitors included) or salicylate with a long half-life (e.g. naproxen, piroxicam, diflusinal, nabumetone, rofecoxib, or celecoxib) it should not be taken 5 days before, the day of, and 2 days after the dose of pemetrexed.
8. Inability or unwillingness to take folic acid, vitamin B12 supplementation, or dexamethasone.
9. Inability to comply with protocol or study procedures.
10. Pregnant or breast-feeding women and childbearing potential women with either a positive or no pregnancy test within 48 hours of the start of treatment. Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
radiological response rate | Three to four weeks after the second cycle of neoadjuvant chemotherapy
  Three to four weeks after the first cycle of neoadjuvant chemotherapy, the same radiological examination as baseline chest CT or PET/CT scans are repeated for tumor response evaluation. Radiographic response was recorded by RECIST 1.1.

SECONDARY OUTCOMES:
Number of Adverse Events of chemotherapy | ten months after neoadjuvant chemotherapy
  1) death due to cancer, toxicity or comorbidity,and 2) toxicity events including Grade 4 neutropenia >7 days; febrile grade 3/4 neutropenia; grade 4 thrombocytopenia >7 days or any grade with bleeding; grade 3/4 nonhematologic toxicity related to chemotherapy (except nausea/vomiting/hair loss)

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan Chen, M.D, PH.D, Study Chair — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided